CLINICAL TRIAL: NCT05706324
Title: A Single-arm, Open-label Phase I Clinical Study to Evaluate the Safety, Tolerability and Immunogenicity of Recombinant COVID-19 Vaccine (Adenovirus Vector) for Inhalation in People 21 to 65 Years Old (Previously Primed With Authorized Vaccines)
Brief Title: Phase Ⅰ Clinical Trial of a Candidate COVID-19 Vaccine
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuhan BravoVax Co., Ltd. (Industry)
Collaborators: National University Hospital, Singapore (Other); Shanghai BravoBio Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BV-C315A-I-2022004
Record Dates: First submitted 2023-01-29; First posted 2023-01-31 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2022-11

CONDITIONS: COVID-19
Keywords: Inhalation; COVID-19 Vaccine
MeSH Terms: conditions — COVID-19; Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): 21~65 year old healthy subjects, received low dose of RCVi
  Interventions: Biological: Recombinant COVID-19 Vaccine (chimpanzee adenovirus vector) for Inhalation
- Medium dose (Experimental): 21~65 year old healthy subjects, received medium dose of RCVi
  Interventions: Biological: Recombinant COVID-19 Vaccine (chimpanzee adenovirus vector) for Inhalation
- High dose (Experimental): 21~65 year old healthy subjects, received high dose of RCVi
  Interventions: Biological: Recombinant COVID-19 Vaccine (chimpanzee adenovirus vector) for Inhalation

INTERVENTIONS:
Biological: Recombinant COVID-19 Vaccine (chimpanzee adenovirus vector) for Inhalation — 0.2mL/dose, Inhalation using a nebulizer
  Other Names: RCVi

SUMMARY:
In this trial, a single-arm, open-label study design will be used to evaluate the safety and tolerability after vaccination with escalating doses of the investigational vaccine (Recombinant COVID-19 Vaccine (chimpanzee adenovirus vector) for Inhalation, RCVi) at low, medium, and high doses in healthy adults (previously primed with authorized vaccines).

ELIGIBILITY:
Inclusion Criteria:

* People aged 21 to 65 years old, with body weight ≥ 50 kg for males and ≥ 45 kg for females, body mass index (BMI) within the range of 19.0-30.0 (including the boundary value), who can provide legal identification;
* Subjects who agree to participate in this study voluntarily and sign an Informed Consent Form.
* Subject who has the ability to understand the study procedures and be able to attend all scheduled follow-up;
* Individuals who completed basic vaccination of licensed vaccine or further received the first booster dose vaccination 4~12 months prior to recruitment in this study（including but not limited to mRNA or non-mRNA vaccine）.
* Female subjects who are not pregnant or breast-feeding;
* Women of childbearing age who agree to use effective contraception during the study; or have been using effective contraception within 2 weeks prior to enrollment.

Exclusion Criteria:

* Those who had fever (body temperature≥ 38.0 °C/100.4 °F), dry cough, fatigue, nasal congestion, runny nose, sore throat, myalgia, diarrhea, shortness of breath, and dyspnea in the past 14 days before vaccination;
* Subject whose SARS-CoV-2 nucleic acid test result is positive;
* Subject with a body temperature of ≥ 38.0 °C/100.4 °F (axillary temperature) on the day of enrollment;
* Subject who has oral ulcers, throat swelling and other oral and nasopharyngeal diseases;
* Subject with abnormal vital signs, physical examination and laboratory test indicators at screening that are judged by clinicians to be clinically significant;
* Subject who has a previous history of severe allergy to any drug, food or vaccination, such as urticaria, anaphylactic shock, allergic laryngeal edema, allergic dyspnea, skin eczema, Henoch-Schonlein purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc.;
* Subject who has suffered from acute disease or in the acute attack stage of chronic disease within 3 days before vaccination, or has used antipyretic, analgesic and anti-allergy drugs;
* Subject within 6 months prior to vaccination participation in a coronavirus (MERS-CoV, SARS-CoV-2) vaccine and/or drug (small molecule) and/or antibody study; Participation in any clinical study within 3 months prior to vaccination or planned participation in other (drug or vaccine) clinical studies during the study;
* Subject who has received other vaccines within 1 month before vaccination;
* Subject who has used immunoenhancers or immunosuppressants in the past 3 months;
* Subject who was diagnosed with congenital or acquired immunodeficiency, or suspected to have systemic diseases that may interfere with the conduct or completion of the study, such as tuberculosis, hepatitis B, hepatitis C, human immunodeficiency virus (HIV), syphilis infection, etc.;
* Subject who was diagnosed with serious diseases, congenital anomalies or chronic disease that may interfere with the conduct or completion of the study (including but not limited to: allergy to vaccines, asthma and other respiratory diseases or chronic bronchitis, hypertension, hypotension, heart disease, kidney disease, diabetes mellitus (type 1 or type 2), autoimmune diseases, thalassemia, malignant tumor, atopy, existing skin diseases, etc.);
* Subject who has received blood or blood-related products (such as blood transfusion, use of human albumin, human immunoglobulin, etc.) within the past 6 months;
* Subject with a history or family history of convulsions, epilepsy, encephalopathy and psychosis;
* Subject with functional asplenia or splenectomy caused by any situation;
* Subject who has any condition that, in the opinion of the investigator, may interfere with the evaluation of the objectives of the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Safety in terms of adverse events | within 30 minutes after vaccination
  Number of Participants with any local and systemic Adverse Events (AEs)
Safety in terms of solicited AEs | within 7 days after vaccination
  Number of Participants with solicited AEs
Safety in terms of unsolicited AEs | within 28 days after vaccination
  Number of Participants with unsolicited AEs
Safety in terms of laboratory-based AEs | 4 days after vaccination
  Changes in laboratory test indicators of clinical significance after vaccination as compared with those before vaccination
Safety in terms of SAEs | within 6 months after vaccination
  Number of Participants with SAEs
Safety in terms of MAAEs and AESIs | within 6 months after vaccination
  Incidence of all Medical Attended Adverse Events (MAAEs) requiring medical attention and Adverse Events of Special Interest (AESIs)

SECONDARY OUTCOMES:
Immunogenicity in terms of Humoral immune response by ELISA | 15, 29 days, 3 and 6 months after vaccination
  GMT of S protein specific antibody by ELISA
Immunogencity in terms of Nab | 15, 29 days, 3 and 6 months after vaccination
  GMT, seroconversion rate and GMFI of neutralizing antibody (NAb) response
Immunogencity in terms of Cellular immune response | 15 days after vaccination
  Intracellular cytokine levels (ICS) in T lymphocytes
Immunogencity in terms of Mucosal immune response | 15 days after vaccination
  Anti-SARS-CoV-2 S protein mucosal IgA antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore